CLINICAL TRIAL: NCT05895682
Title: A Clinical Trial to Verify the Accuracy of Seers Technology's Pulse Oximeter (mobiCARE +Pulse, MP100W) in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seers Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-1657
Record Dates: First submitted 2023-05-21; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Oxygen Saturation
Keywords: Oxygen Saturation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induced hypoxia (Experimental): Volunteers were monitored using end-tidal carbon dioxide partial pressure and fraction of inspired oxygen. Each volunteer was placed in a semi-Fowler's position and connected to a breathing circuit to administer the nitrogen-air-carbon dioxide mixtures. A nose clip was applied to prevent breathing of room air. For frequent blood sampling, an arterial cannula was placed in the radial artery of each volunteer. Pulse oximeter probes were simultaneously attached to each volunteer's fingers. Each volunteer was exposed to various levels of induced hypoxia from 70~100% of SaO2. Each plateau of oxygen saturation was maintained for at least 30 s until stabilization, after which 1 ml of arterial blood was drawn into a heparinized syringe. The study period consisted of two rounds of hypoxia, and the volunteers were maintained on room air between each round. SaO2 measurements using a CO-oximeter were used as a reference for the SpO2 accuracy.
  Interventions: Device: mobiCARE +Pulse (MP100W)

INTERVENTIONS:
Device: mobiCARE +Pulse (MP100W) — Volunteers were monitored using end-tidal carbon dioxide partial pressure and fraction of inspired oxygen. Each volunteer was placed in a semi-Fowler's position and connected to a breathing circuit to administer the nitrogen-air-carbon dioxide mixtures. A nose clip was applied to prevent breathing of room air. For frequent blood sampling, an arterial cannula was placed in the radial artery of each volunteer. Pulse oximeter probes were simultaneously attached to each volunteer's fingers. Each volunteer was exposed to various levels of induced hypoxia from 70~100% of SaO2. Each plateau of oxygen saturation was maintained for at least 30 s until stabilization, after which 1 ml of arterial blood was drawn into a heparinized syringe. The study period consisted of two rounds of hypoxia, and the volunteers were maintained on room air between each round. SaO2 measurements using a CO-oximeter were used as a reference for the SpO2 accuracy.

SUMMARY:
It is important to evaluate the accuracy of the pulse oximeter, which is commonly used in clinical practice. The US FDA only allows the use of devices that meet the ISO 80601-2-61:2017 standard in the United States. According to the ISO 80601-2-61:2017 standard, the accuracy of the oxygen saturation (SpO2) of the pulse oximeter should have an error range of less than 4.0% compared to the actual arterial blood oxygen saturation (SaO2) in the range of 70-100%. To prove compliance with this requirement, it is necessary to conduct a clinical trial that induces hypoxemia in healthy adults and compares and evaluates the arterial blood oxygen saturation values of the pulse oximeter's SpO2 and the arterial blood oxygen saturation values of the carbon monoxide-oxygen meter (CO-oximeter).

ELIGIBILITY:
Inclusion Criteria:

* healthy adults between 20 and 50 years
* volunteers who have plasma proportion of carboxyhemoglobin 3%
* volunteers who have plasma proportion of methemoglobin 2%
* volunteers who have total plasma hemoglobin concentration over 10 g/dL

Exclusion Criteria:

* History of respiratory diseases
* History of cardiovascular disease
* Smokers (including ex-smokers)
* Pregnant
* History of fainting
* History of diabetes
* Obesity (BMI> 30 kg/m2)
* Allen's test results, those who do not recover the color of their fingers and palms within 10 seconds
* History of allergic reaction to lidocaine, a local anesthetic

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-29 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of SpO2 | 2 day
  The root-mean-square of the difference between the observed pulse oximetry value (SpO2) and the carbon monoxide-oxygenometer arterial blood reference value (SRi) within the range of 70-100% of arterial oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Seers Technology Co., Ltd., Pyeongtaek-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No